CLINICAL TRIAL: NCT04296045
Title: A Randomised, Double-blind, Placebo-controlled, Cross-over Study, to Investigate the Effect of Maize Cob Extract on Post-prandial Glucose and Insulin Responses in Healthy Males
Brief Title: A Study to Investigate the Effect of MCE on Glucose and Insulin Responses in Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Glycoscience (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CG1142
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Dysglycemia
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glucose (Active Comparator): Glucose
  Interventions: Dietary Supplement: Glucose
- MCE (Experimental)
  Interventions: Dietary Supplement: MCE
- MCE + Glucose (Experimental)
  Interventions: Dietary Supplement: MCE; Dietary Supplement: Glucose

INTERVENTIONS:
Dietary Supplement: MCE — Ingestion of 15g MCE in water after min 10 hours of fasting
  Arms: MCE; MCE + Glucose
Dietary Supplement: Glucose — Ingestion of 15g glucose in water after min 10 hours of fasting
  Arms: Glucose; MCE + Glucose

SUMMARY:
Maize Cob Extract (MCE) is intended to be used as a bulking agent in food. The purpose of this study is to determine the glycaemic and insulinemic response of MCE consumed in isolation compared to glucose; the glycaemic and insulinemic response will also be determined for MCE alone and in combination with glucose. This is a randomised, double-blind, single-centre trial in 10 healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent;
* Be between 18 and 60 years of age inclusive;
* Have a body mass index <30 Kg/m2;
* Have a fasting glucose level of ≤6.0 mmol/L
* Be in general good health, as determined by the investigator;
* Be willing to fast for at least 10 hours before the study visit.

Exclusion Criteria:

* The presence of any of the following criteria will exclude the participant from participating in the study:
* Are less than 18 or greater than 60 years of age;
* Recent gastroenteritis or food borne illness such as confirmed food poisoning within the past 4 weeks;
* Have taken a medication or dietary supplement that may influence GI activity within the 2-weeks prior to screening;
* Have a history of abdominal surgery (excluding appendectomy);
* Have taken anaesthesia within the past 4 weeks;
* Have taken antibiotics within the past 12-weeks;
* Have a recent history of drug and/or alcohol abuse at the time of enrolment;
* Are a smoker (defined as >5 cigarettes/week);
* Have made any major dietary change in the past 3 months;
* Have planned major changes in lifestyle (i.e. diet, dieting, exercise level, travelling) during the duration of the study;
* Have an active gastrointestinal disorder or previous gastrointestinal surgery;
* Have irritable bowel syndrome, diagnosed or undiagnosed and treated with chronic medications;
* Have a metabolic or endocrine disorder such as diabetes, thyroidism, or other metabolic disorder;
* Have a severe chronic disease i.e. cancer, renal failure, hepatitis, HIV, cirrhosis etc., or with a history of such diseases;
* Have a gastrointestinal disease i.e., chronic diarrhoea, Crohn's disease, ulcerative colitis, diverticulosis, stomach or duodenal ulcers, or with a history of such diseases;
* Are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a systemic steroid for >30 days, or chemotherapy or radiotherapy within the last year);
* Experiences alarm features such as weight loss, rectal bleeding, recent change in bowel habit (<3 months) or abdominal pain;
* Participants who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial;
* Participant is currently receiving treatment involving experimental drugs. If the participant has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Difference in venous glucose from incremental area under the curve (iAUC) (T-15 to T120 minutes) | Through intervention periods of two hours

SECONDARY OUTCOMES:
Difference in venous insulin from incremental area under the curve (iAUC) (T-15 to T120 minutes) | Through intervention periods of two hours
Maximal concentrations for glucose and insulin (Cmax) | Through intervention periods of two hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nicholson, M.Phil; M.Sc, Study Director — Cambridge Glycoscience; Timothy Dinan, M.D; Ph.D; D.Sc, Principal Investigator — Atlantia Food Clinical Trials
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided